CLINICAL TRIAL: NCT04788056
Title: Parasternal Subpectoral Plane Blocks for Patients Undergoing Cardiac Surgery Involving Median Sternotomy - a Study of Opioid and Pain Reduction
Brief Title: Parasternal Subpectoral Plane Blocks for Cardiac Surgery Via a Midline Sternotomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no support received
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kamen Vlassakov, Director of Regional Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P000486
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Saline and Bupivacaine are both clear fluids and look identical. Research pharmacy will prepare blinded solutions for use in study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Experimental): PSPB catheters will be placed with 60mL of 0.2% bupivacaine and continue to infuse bupivacaine 0.125% at 10mL/hr through the catheter
  Interventions: Procedure: Parasternal Subpectoral Plane Block
- Saline (Placebo Comparator): PSPB catheters will be placed with 60mL of saline and continue to infuse saline through the catheters.
  Interventions: Procedure: Parasternal Subpectoral Plane Block

INTERVENTIONS:
Procedure: Parasternal Subpectoral Plane Block — Nerve block catheter inserted into plane between rib cartilages and pectoralis muscle.

SUMMARY:
To better determine whether parasternal subpectoral plane blocks (PSPB) infusing bupivacaine for midline sternotomy decreases opioid consumption and pain scores.

This is a prospective, blinded randomized controlled trial with 2 arms. 1 arm is the saline control arm, PSPB catheters will be placed with saline and continue to infuse saline. The other arm is bupivacaine study arm, PSPB catheters will be placed with bupivacaine and continue to infuse the local anesthetic.

DETAILED DESCRIPTION:
Subjects will be randomized to receive PSPB catheters infusing either bupivacaine or saline. Randomization will be achieved using a computer-generated randomization scheme. The surgeon, nurse, anesthetist and patient will be blinded. The investigational drug service will prepare blinded solutions (bupivacaine 0.2% or saline syringes) for performance of the block. They will also prepare bags (either bupivacaine 0.125% or saline) to be infused through the catheter.

Following skin closure, but before removal of the surgical drapes, regional anesthesiologists will scrub in, gown and perform the placement of PSPB catheters under strict surgical aseptic technique. Real-time ultrasound (US) imaging will be used to visualize the pectoralis major muscle and its corresponding rib cartilages, and a needle/introducer sheath will be guided parasternally into the fascial plane. The needle will be advanced in the plane, hydro-dissecting with 30 mL of bupivacaine 0.2% in the study group or 30 mL of saline in the control group per side. Following hydro-dissection, a 5 in. multiport catheter will be inserted via the sheath, and the catheter will be secured following US confirmation of appropriate catheter position. This procedure will then be repeated on the other side. After completion of bilateral PSPB catheters, patients will remain intubated and be transferred to the CSICU on a sedation regimen at the discretion of the intraoperative anesthesia team. Upon dropping off to the ICU, each catheter will be attached to a programmable pump infusing plain bupivacaine 0.125% at 10 mL/hr or saline infusing at 10 mL/hr. Once again, the solution to be infused postoperatively will be prepared by pharmacy and blinded from the patient, nurse, and postoperative pain service providers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Aged 18 - 80 years
3. scheduled for primary elective cardiac surgery via median sternotomy
4. willingness to undergo psychosocial testing
5. willingness to participate in long-term follow up
6. willingness to be randomized to receive local anesthetic or saline infusion through PSPB catheters
7. access to an email and computer

Exclusion Criteria:

1. Allergy to opioids
2. allergy to bupivacaine
3. emergency surgery
4. unable to provide informed consent
5. weight less than 50kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | 2 days
  Cumulative opioid consumption on post-operative day 1 and 2

SECONDARY OUTCOMES:
Acute Postoperative Pain scores | through initial hospital stay, an average of 5 days
  At rest and activity, on a numerical rating scale (NRS) 0-10
Persistent Postoperative Pain scores | Measured at 1 year
  Persistent midline sternotomy pain, on a numerical rating scale (NRS) 0-10
Pain and patient characteristics | 1 year
  Whether there is a correlation between development of persistent post-sternotomy pain and psychosocial/psychophysical characteristics. Will be ascertained from a variety of questionnaires (i.e. brief pain index, brief symptom inventory, coping strategies, fibromyalgianess, pain catastrophizing scale, positive and negative affect scale, PROMIS anxiety short form (SF), PROMIS depression SF, PROMIS sleep disturbance SF
Incidence of arrhythmia | Hospital stay, an average of 5 days
  Whether active bupivacaine group has lower incidence of arrythmia versus saline control group. And whether this correlates to a certain plasma bupivacine level
Time to extubation | Post-operative day 1
  From arrival time to ICU to extubation
Length of ICU stay | From arrival to ICU to discharge to floor, up to 5 days
  When patients are deemed ready to be discharged from ICU
Length of hospital stay | From arrival to ICU to discharge from hospital, up to 5 days
  When patients are deemed ready to be discharged from hospital
Incidence of delirium | Time in ICU to discharge to floor, up to 3 days
  Assessed using CAM-ICU
Time to first opioid administration after extubation | Extubation to first opioid administration, up to 3 days
  When patient first requests opioid after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Kamen Vlassakov, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] Edwards RR, Cahalan C, Mensing G, Smith M, Haythornthwaite JA. Pain, catastrophizing, and depression in the rheumatic diseases. Nat Rev Rheumatol. 2011 Apr;7(4):216-24. doi: 10.1038/nrrheum.2011.2. Epub 2011 Feb 1. PMID 21283147
- [Background] Taillefer MC, Carrier M, Belisle S, Levesque S, Lanctot H, Boisvert AM, Choiniere M. Prevalence, characteristics, and predictors of chronic nonanginal postoperative pain after a cardiac operation: a cross-sectional study. J Thorac Cardiovasc Surg. 2006 Jun;131(6):1274-80. doi: 10.1016/j.jtcvs.2006.02.001. PMID 16733157